CLINICAL TRIAL: NCT07085260
Title: Time-series Changes in Optic Nerve Sheath Diameter and Its Association With Treatment Response After Epidural Blood Patch in Patients With Spontaneous Intracranial Hypotension
Brief Title: ONSD Changes and Treatment Response After Epidural Blood Patch in Spontaneous Intracranial Hypotension
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2025-0662
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Spontaneous Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"This is a prospective observational study investigating changes in optic nerve sheath diameter (ONSD) and its association with clinical improvement following epidural blood patch (EBP) in patients with spontaneous intracranial hypotension (SIH). SIH is a secondary headache disorder caused by cerebrospinal fluid (CSF) leakage or low CSF pressure and is often underdiagnosed due to its diverse and nonspecific presentation.

ONSD, measured via ocular ultrasonography, has emerged as a non-invasive surrogate marker for intracranial pressure (ICP), with its diameter decreasing in states of intracranial hypotension. Prior studies suggest that posture-related ONSD differences (e.g., between supine and upright positions) may be more sensitive in SIH than static values alone, and that ONSD may increase following dural repair, correlating with symptom improvement. However, no studies to date have systematically examined the time-series evolution of ONSD around EBP in SIH patients.

In this study, adult patients diagnosed with SIH and scheduled for their first EBP at our hospital will be enrolled. ONSD will be measured using standardized ultrasound protocols at three timepoints: immediately before EBP (T0), immediately after EBP (T1), and at follow-up admission two weeks later (T2). Measurements will be taken in both supine and upright positions at each timepoint to calculate posture-related changes (ΔONSD = supine - upright).

Concurrently, clinical symptom assessments will be conducted using standardized instruments: Numeric Rating Scale (NRS) for headache intensity, HIT-6 for headache impact, PHQ-9 and GAD-7 for emotional distress, and EQ-5D-5L for quality of life. These will be administered at T0 and T2.

Primary outcomes include the change in ΔONSD over time. Secondary outcomes involve the correlation between ΔONSD and clinical improvement metrics (e.g., reduction in NRS or HIT-6 scores). Descriptive and inferential statistics will be performed, including repeated measures ANOVA or Friedman test for time-series data, and Pearson or Spearman correlation for association analysis.

All ONSD measurements and EBP procedures will be performed by the same experienced anesthesiologist following a standardized institutional protocol. This study aims to evaluate whether ONSD can serve as a quantitative imaging biomarker reflecting treatment responsiveness in SIH.

ELIGIBILITY:
Inclusion Criteria:

* dults aged 19 years or older diagnosed with spontaneous intracranial hypotension (SIH) according to the 3rd edition of the International Classification of Headache Disorders (ICHD-3), and scheduled to undergo their first epidural blood patch (EBP) at our institution.

Individuals who have received sufficient explanation of the study purpose and procedures, and voluntarily provided written informed consent with full legal capacity.

Exclusion Criteria:

* Patients younger than 19 years. Patients with secondary headache clearly attributable to other causes such as trauma, medications, or infections.

Individuals who are unable or unwilling to voluntarily provide informed consent for study participation.

Patients with cognitive impairment, psychiatric disorders, or language difficulties that interfere with completing questionnaires or clinical assessments.

Patients with medical contraindications to EBP, such as active infection or bleeding tendency.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include adults aged ≥19 years who are scheduled to receive their first epidural blood patch (EBP) at Severance Hospital for clinically diagnosed spontaneous intracranial hypotension (SIH), based on the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria by the International Headache Society. Only patients who voluntarily provide written informed consent after receiving sufficient explanation about the study's objectives and procedures will be enrolled. All participants must be legally capable of providing consent.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Change in Optic Nerve Sheath Diameter (ΔONSD) across three time points | Baseline (pre-EBP)
  Measurement of optic nerve sheath diameter (ONSD) in both supine and upright positions using standardized ocular ultrasonography at three time points. The primary variable is ΔONSD (supine - upright), and the primary outcome is the time-series change of ΔONSD after epidural blood patch (EBP) treatment in patients with spontaneous intracranial hypotension (SIH). Changes will be analyzed using repeated measures ANOVA or nonparametric equivalents depending on distribution.
Change in Optic Nerve Sheath Diameter (ΔONSD) across three time points | immediate post-EBP (within 1 hour)
  Measurement of optic nerve sheath diameter (ONSD) in both supine and upright positions using standardized ocular ultrasonography at three time points. The primary variable is ΔONSD (supine - upright), and the primary outcome is the time-series change of ΔONSD after epidural blood patch (EBP) treatment in patients with spontaneous intracranial hypotension (SIH). Changes will be analyzed using repeated measures ANOVA or nonparametric equivalents depending on distribution.
Change in Optic Nerve Sheath Diameter (ΔONSD) across three time points | 2 weeks post-EBP
  Measurement of optic nerve sheath diameter (ONSD) in both supine and upright positions using standardized ocular ultrasonography at three time points. The primary variable is ΔONSD (supine - upright), and the primary outcome is the time-series change of ΔONSD after epidural blood patch (EBP) treatment in patients with spontaneous intracranial hypotension (SIH). Changes will be analyzed using repeated measures ANOVA or nonparametric equivalents depending on distribution.

SECONDARY OUTCOMES:
Correlation between changes in ΔONSD and clinical symptom improvement | Baseline and 2 weeks post-EBP
  To evaluate the association between ΔONSD change and changes in clinical assessment scores, including Numeric Rating Scale (NRS), Headache Impact Test-6 (HIT-6), Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), and EQ-5D-5L. Correlation analysis (Pearson or Spearman) will be performed based on data distribution.

IPD SHARING:
Plan to Share IPD: Undecided